CLINICAL TRIAL: NCT02001545
Title: REal World Information on Cardiovascular Drug Management Patterns in Acute Coronary Syndrome paTients
Acronym: RE-ACT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CBG-XXX-2013/1
Record Dates: First submitted 2013-11-18; First posted 2013-12-05 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndrome, antithrombotic management patterns,quality of life, acute clinical management strategies
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with STEMI and NSTEMI: Patients aged 18 years or older, hospitalized and diagnosed with STEMI (ST-segment elevation myocardial infarction) or NSTEMI (non-ST-segment elevation myocardial infarction) within 24 hours of symptom onset.

SUMMARY:
RE-ACT is a national, multi-centre, observational, prospective, longitudinal cohort study which will include patients hospitalized for ACS within 24 hours of symptom onset and who have a final diagnosis of ST-segment elevation myocardial infarction (STEMI) or non-ST-segment elevation myocardial infarction (NSTEMI). This study aims to describe the short-term (at the end of the first month after index event) antithrombotic management patterns in a "real-life" setting for patients hospitalized with an acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Provision of subject informed consent
* Patients hospitalized and diagnosed with STEMI or NSTEMI
* Hospitalized within 24 hours of onset of symptoms or transferred from another hospital within 24 hours of the onset of symptoms

Exclusion Criteria:

* STEMI and NSTEMI precipitated by or as a complication of surgery, trauma, or GI bleeding or post-PCI.
* STEMI and NSTEMI occurring in patients already hospitalized for other reasons.
* Presence of any condition/circumstance which in the opinion of the investigator could significantly limit the complete follow up of the patient (e.g. tourist, non-native speaker or does not understand the local language, psychiatric disturbances).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older, hospitalized and diagnosed with STEMI (ST-segment elevation myocardial infarction) or NSTEMI (non-ST-segment elevation myocardial infarction) within 24 hours of symptom onset.
Sampling Method: Probability Sample
Enrollment: 814 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Short-term antithrombotic management patterns (AMPs) in a real-life setting for patients hospitalized with an ACS | Baseline
  Descriptive statistics will be calculated for this outcome measure using frequency tables (n, frequency and percentage). Antithrombotic management patterns will be grouped taking into account only the different treatment options shown by the descriptive analysis.

SECONDARY OUTCOMES:
Variations in the acute clinical management strategies and AMPs. | Baseline
  Descriptive statistics will be calculated for this outcome measure using frequency tables (n, frequency and percentage).
Impact of the different AMPs on quality of life at discharge from hospital (using EuroQoL-5D). | Baseline
  Descriptive statistics will be calculated for this outcome measure using frequency tables (n, mean, median, standard deviation, minimum and maximum)
Impact of the different AMPs on quality of life at the end of the first month after discharge from the hospital (using EuroQoL-5D). | At the end of the first month after index event
  Descriptive statistics will be calculated for this outcome measure using frequency tables (n, mean, median, standard deviation, minimum and maximum)
Determinants of AMP choices (i.e. patient's characteristics, hospital characteristics, coronary intervention strategies and type of coronary stents used) | Baseline
  Descriptive statistics will be calculated for this outcome measure using frequency tables (n, frequency and percentage).

CONTACTS AND LOCATIONS:
Overall Officials: Elina Trendafilova, Ass. Prof. M.D, Principal Investigator — National Cardiology Hospital, Sofia; Vasil Velchev, Ass. Prof. M.D., Principal Investigator — University Hospital St. Anna
Locations (8):
- Bulgaria (8):
  - Research Site, Blagoevgrad
  - Research Site, Burgas
  - Research Site, Lovech
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Vratsa